CLINICAL TRIAL: NCT00925678
Title: A Double-blind, Placebo-controlled, Randomised Study to Investigate the Tolerability, Safety, Pharmacokinetics and Pharmacodynamics of Single Ascending Doses of DSP-3025 Administered Intranasally to Healthy Male Volunteers and Seasonal Allergic Rhinitis Male Patients Out of Season
Brief Title: DSP-3025 Study of Healthy Male Volunteers and Seasonal Allergic Rhinitis Male Patients Out of Season
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double
Other Study IDs: D7002013
Record Dates: First submitted 2009-06-19; First posted 2009-06-22 (Estimated); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Allergic Rhinitis; Healthy Volunteer
MeSH Terms: conditions — Rhinitis, Allergic

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: DSP-3025
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: DSP-3025
  Arms: 1
Drug: Placebo
  Arms: 2

SUMMARY:
Investigate safety/tolerability after a single dose intranasal administration of DSP-3025 comparator placebo to healthy male volunteers and seasonal allergic rhinitis male patients out of season.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.5 and 25 kg/ m2 and a weight between 50 and 80 kg
* No clinically relevant abnormal findings
* History of cedar and/or Japanese cypress pollen induced seasonal allergic rhinitis for at least the previous 2 years (only Allergic rhinitis)

Exclusion Criteria:

* Acute illness which requires medical intervention
* Definite or suspected personal history of adverse drug reactions or drug hypersensitivity
* Clinical relevant disease or disorder (past or present)
* A history of asthma

Ages: 20 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2009-06

PRIMARY OUTCOMES:
Incidence/nature of adverse events, 12-lead ECG, pulse, BP, body temperature, spirometry

SECONDARY OUTCOMES:
Clinical chemistry, haematology, urinalysis
Nasal symptoms and peak nasal inspiratory flow
Pharmacokinetics
Biomarkers nasal lavage and blood

CONTACTS AND LOCATIONS:
Locations (1):
- Kitasato University East Hospital, Sagamihara, Kanagawa, Japan